CLINICAL TRIAL: NCT00299429
Title: Randomised Comparison of Minimally Invasive Direct Coronary Artery Bypass Grafting and Percutaneous Coronary Intervention With Drug-eluting Stents in Patients With Proximal Stenosis of the Left Anterior Descending Coronary Artery
Brief Title: MIDCAB Versus DES in Proximal LAD Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Cordis Medizinische Apparate GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-Thiele
Record Dates: First submitted 2005-09-09; First posted 2006-03-06 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2007-03

CONDITIONS: Coronary Artery Disease
Keywords: Stent; drug-eluting stent; Minimally invasive bypass surgery; left anterior descending
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIDCAB Surgery (Active Comparator): MIDCAB Surgery
  Interventions: Procedure: Stenting and minimally invasive bypass surgery
- PCI with drug-eluting stent (Experimental): PCI with DES
  Interventions: Procedure: PCI with DES

INTERVENTIONS:
Procedure: Stenting and minimally invasive bypass surgery
  Arms: MIDCAB Surgery
Procedure: PCI with DES — PCI with DES
  Arms: PCI with drug-eluting stent

SUMMARY:
Percutaneous coronary intervention with a sirolimus-coated stent compared to minimally invasive bypass surgery in patients with isolated proximal left anterior descending coronary arteries in terms of non-inferiority of an end point combining mortality, acute myocardial infarction and rate of reintervention of the target vessel within one year.

ELIGIBILITY:
Inclusion Criteria:

1. Single-vessel disease of the proximal LAD with a stenosis > 50% (multivessel disease only if further coronary vessel stenoses do not require treatment)
2. Patients with angina pectoris (CCS 1-4)
3. Asymptomatic patients if clear signs of ischemia in the segments supplied by the LAD as assessed by bicycle ergometry or treadmill and/or scintigraphically and/or stress echo
4. Patients for whom both methods of treatment are equally possible
5. Consensus between the cardiac surgeon and the cardiologist that both inclusion and exclusion criteria are met in the selected case
6. Informed consent of the patient.

Exclusion Criteria:

1. Patients < 18 years
2. Pregnancy
3. Previous coronary artery bypass surgery
4. Concomitant diseases that lead to a greater risk for each of the treatment strategies
5. Significant peripheral arterial occlusive disease
6. Concomitant disease with limited life expectancy (e.g. malignant tumours that have not been curatively treated)
7. Objective follow-up examination not possible due to physical or mental handicap
8. Participation in another study.

Angiographical exclusion criteria:

1. Left main stem stenosis
2. Multivessel disease for which surgical or interventional therapy on other vessel areas is required.
3. Diagonal/septal branch > 1.5 mm, which might be compromised by a stent
4. Need for acute intervention (e.g. acute myocardial infarction)
5. Total occlusion of the LAD

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 12 months

SECONDARY OUTCOMES:
Perioperative complications | 30 days
CCS-Classification | 12 months
cost-effectiveness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] Blazek S, Rossbach C, Borger MA, Fuernau G, Desch S, Eitel I, Stiermaier T, Lurz P, Holzhey D, Schuler G, Mohr FW, Thiele H. Comparison of sirolimus-eluting stenting with minimally invasive bypass surgery for stenosis of the left anterior descending coronary artery: 7-year follow-up of a randomized trial. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):30-8. doi: 10.1016/j.jcin.2014.08.006. Epub 2014 Dec 10. PMID 25499302
- [Derived] Thiele H, Neumann-Schniedewind P, Jacobs S, Boudriot E, Walther T, Mohr FW, Schuler G, Falk V. Randomized comparison of minimally invasive direct coronary artery bypass surgery versus sirolimus-eluting stenting in isolated proximal left anterior descending coronary artery stenosis. J Am Coll Cardiol. 2009 Jun 23;53(25):2324-31. doi: 10.1016/j.jacc.2009.03.032. PMID 19539141